CLINICAL TRIAL: NCT06262867
Title: Pragmatic, Randomized, Controlled Trial of Early Cow's Milk, Egg, and Peanut Allergen Introduction and Maintenance in Healthy and High-Risk Infants
Brief Title: Early Allergen System Experience
Acronym: EASE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prollergy dba Ready Set Food (Other)
Collaborators: ObvioHealth (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ReadySetFood
Record Dates: First submitted 2024-01-26; First posted 2024-02-16 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-02

CONDITIONS: Food Allergy in Infants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants randomized to the intervention group will receive an early allergen introduction supplement.
  Interventions: Dietary Supplement: Ready. Set. Food! Stage 1 Mix ins
- Control (No Intervention): Participants randomized to the control group will follow the guidance of their pediatrician.

INTERVENTIONS:
Dietary Supplement: Ready. Set. Food! Stage 1 Mix ins — These supplements contain cow's milk, eggs, and peanuts.
  Other Names: Ready. Set. Food! Stage 2 Mix ins
  Arms: Intervention

SUMMARY:
Multiple clinical trials have demonstrated that early allergen introduction, feeding babies common food allergens before six months, decreases children's risk of developing a food allergy. Despite successful food allergy introduction trials showing that food allergies can be prevented, early introduction in the required amount can be challenging for parents. In some studies, less than 20% of parents introduce peanuts before their child is six months old, and few feed them regularly after introduction. Ready. Set. Food! is a direct-to-consumer product that offers a convenient supplement with a daily dose regimen that can be added to breastmilk, formula, or food to make early allergen introduction easy. The formulation includes cow's milk, egg, and peanut, representing the majority of childhood food allergies, and the protein levels are based on doses found to be effective in clinical trials. Over 200,000 infants have used Ready. Set. Food!.

This study investigates the effectiveness of introducing common allergens to infants with the goal of preventing food allergies. The study will enroll 1,100 infants stratified by their risk of developing a food allergy who are assigned to either receive Ready. Set. Food! supplements or follow standard allergen introduction practices recommended by their pediatrician.

The goal of this study is to assess how Ready. Set. Food! allergen introduction supplements improve the experience of parents introducing allergens, decrease healthcare costs related to food allergies, and decrease food allergy prevalence.

DETAILED DESCRIPTION:
Childhood food allergy is characterized by the loss of immune tolerance to specific foods, triggering immune reactions that manifest in various symptoms, including skin, respiratory, gastrointestinal, and cardiovascular issues. Common triggers in children include proteins from cow's milk, hen's egg, peanuts, tree nuts, wheat, soy, and sesame. The prevalence of food allergy has surged, affecting 8% of United States (U.S.) children, with a notable increase in food-induced anaphylactic reactions. Peanut allergy, in particular, tends to be persistent, with a lower resolution rate than egg and cow's milk allergy. Milk and egg allergies are more likely to resolve, but make up the bulk of food allergies in infants and young toddlers and are associated with nutritional deficiencies and growth restriction.

Several randomized, controlled trials have investigated early allergen introduction to prevent food allergy. The Learning Early About Peanut (LEAP) study demonstrated a significant reduction in peanut allergy by introducing peanuts early, irrespective of baseline sensitization. Follow-up indicated sustained risk reduction. The Enquiring About Tolerance (EAT) trial explored the early introduction of multiple allergens, showing a lower relative risk of food allergy, particularly peanut and egg allergy in infants who were regularly fed the allergens. The Prevention of Egg Allergy in High-Risk Infants with Eczema (PETIT) study focused on egg introduction, revealing a preventive effect with gradual, consistent consumption. The Strategy for Prevention of Milk Allergy by Daily Ingestion of Infant Formula in Early Infancy (SPADE) study highlighted that early ingestion of cow's milk formula reduced cow's milk allergy risk. Early Food Intervention and Skin Emollients to Prevent Food Allergy in Young Children (PreventADALL), a multicenter trial, combined skin and food interventions, demonstrating a reduced food allergy at 36 months. Government bodies and professional societies, including National Institute of Allergy and Infectious Disease (NIAID), American Academy of Pediatrics (AAP), American Academy of Allergy, Asthma, and Immunology (AAAAI), American College of Allergy, Asthma, and Immunology (ACAAI), and Canadian Society of Allergy and Clinical Immunology (CSACI), recommend early allergen introduction based on these trials.

Guidelines advise introducing peanut and other allergenic foods by 6 months, avoiding delays, especially for high-risk infants with severe eczema or egg allergy. The PreventADALL trial supported early exposure to allergenic foods to prevent food allergy. The Center for Disease Control (CDC) reported varying ages of complementary food introduction in the U.S., with a prevalence of early introduction before 4 months. Despite guidelines, low adherence rates were observed in the PreventADALL trial.

Safety of Introducing Food to Infants:

Infant anaphylaxis is rare, with allergic infants typically presenting with mild to moderate symptoms. Clinical trials and real-world studies demonstrated low rates of severe reactions, even in higher-risk infants. Recent guidelines focus on early, regular allergen ingestion, emphasizing the safety of introducing potentially allergenic foods to infants.

Study Rationale:

The trials promoting early allergen introduction face challenges in widespread adoption due to the difficulty of maintaining feeding requirements. In the case of LEAP, parents were contacted 104 times throughout the study to ensure compliance. For the EAT study, only 43% of parents could maintain the feeding requirements, which included large amounts of solid foods for infants who had not started eating otherwise, and some had difficulties doing so. Consumption levels were a critical factor for the EAT study: the reduction in food allergy was only shown to be statistically significant in the group of families who could maintain a certain level of compliance. The data from LEAP and EAT indicate that ingestion of 2 grams of protein per week of the allergenic food was required to decrease the risk of food allergy. Ingesting 2 grams of protein per week of allergenic food is crucial. Early introduction, before 6 months, is vital, but a method for infants not developmentally ready for solids is needed.

Ready. Set. Food! Stage 1 and 2 Mix-ins address these challenges with a patented direct-to-consumer product introducing top pediatric allergens in stages. It covers cow's milk, egg, and peanut, representing over 80% of childhood food allergies. The regimen, dissolved in a bottle of breast milk or formula, follows a sequential introduction process, replicating home food introduction. The formulation aims to promote tolerance development via the gastrointestinal system, aligning with prevention trials. Over 150,000 infants have used Ready. Set. Food! and in preliminary assessments of consumers, more than 95% achieved the clinically recommended duration with very few allergic reactions.

The study design was created to mimic the real-world environment in which caregivers would introduce allergens to their infants. Therefore, the study design avoids in-person visits with the study team and prescriptive requirements for testing and evaluation. Due to the nature of the study, blinding the interventional group would not replicate a real-world environment. In addition, an unblinded study allows caregivers to seek additional information and support, such as they would in a real-world environment, and make decisions based on the early allergen introduction they have completed.

ELIGIBILITY:
Inclusion Criteria:

* Full term, singleton birth
* Infant will be 2-5 months old at the time of study enrollment
* Able to participate in the study under the supervision of a caregiver or legal guardian -who must be:

  1. At least 18 years of age
  2. The caregiver or legal guardian of the infant
  3. Living with the infant for the duration of the study
  4. Willing to follow all caregiver responsibilities
  5. Willing and able to sign the electronic Informed Consent
  6. Willing to conform to all protocol requirements (e.g., completion of study questionnaires and procedures, and reporting of AEs)
* Caregiver or legal guardian who owns a functioning smartphone device, has access to an internet connection (Wi-Fi or data plan), and is willing to download the study app

Exclusion Criteria:

* Known sensitivity/allergy to egg, cow's milk, or peanut (including products containing egg, cow's milk, or peanut) or undergoing evaluation for reactions due to cow's milk, egg, or peanut exposure (including exposure to products containing egg, cow's milk, or peanut).
* Participating in a clinical trial and/or treated with any investigational product within 3 months preceding the first dose of study product.
* Clinically significant medical conditions such as cardiac disease or lung disease, and/or babies who have bloody stools that have required milk elimination that are unstable or uncontrolled and may interfere with a participant's participation in the study in the opinion of the medically qualified investigator.
* Other severe, acute or chronic, medical or psychiatric condition(s) or laboratory abnormality(ies) that may increase the risk associated with study participation or intervention product administration or may interfere with the interpretation of study results, and in the judgment of the medically qualified investigator, would make the participant inappropriate for entry into this study.
* Preterm delivery (<37 weeks [259 days] gestational age).
* Admission to the neonatal unit ≥ 3 days for issues other than establishment of normal feeding.
* Chronic use of antibiotics (≥ 28 consecutive days)
* Evidence of a baseline illness that would, in the opinion of the PI, introduce a significant safety concern if the infant is enrolled in the study or otherwise preclude study participation.
* Significant birth defect/complication that would, in the opinion of the PI, create a safety concern or otherwise confound the study (e.g., abdominal wall defects, congenital heart disease).
* Medical condition (infant) that, in the opinion of the PI, may significantly alter gut microbiota or healthy immune responses.
* Maternal infection with human immunodeficiency virus, tuberculosis, hepatitis C, or hepatitis B.
* Caregiver condition that, in the opinion of the PI, would not allow the Caregiver and/or infant to comply with the study protocol requirements.
* History of immunocompromised conditions. Is related to persons involved directly or indirectly with the conduct of this study (i.e., PI, sub-investigators, study coordinators, other study personnel, employees of Ready. Set. Food! contractors of Ready. Set. Food! and the families of each).

Ages: 2 Months to 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1110 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of caregivers who are adherent with the evidence-based guidance for cow's milk, egg, and peanut during the 6 - month period | 6 months of intervention
  Adherence will be measured using a food frequency questionnaire

SECONDARY OUTCOMES:
Frequency of caregiver-reported allergy or food introduction-related adverse events (AEs) after introduction of cow's milk, egg, and peanut | 12 months of age
  AEs will be evaluated by study PI
Frequency of caregiver-reported serious adverse events (SAEs) after introduction of cow's milk, egg, and peanut | 12 months of age
  SAEs will be evaluated by study PI
Frequency of caregiver-reported special interest adverse events (FPIES and anaphylaxis) after introduction to cow's milk, egg, and peanut by 12 months of age | 12 months of age
  AEs of special interest will be evaluated by study PI

OTHER OUTCOMES:
The proportion of caregivers who are satisfied with introduction of egg, cow's milk, and peanut | 12 months of age
  Assessed by parental report
The total allergy-related healthcare costs | 24 months of age
  Assessed by claims evaluation
The proportion of participants with food allergy to cow's milk, egg, or peanut | 24 months of age
  Documented by a diagnosis code in claims data
The proportion of participants with a suspected food allergy | 24 months of age
  Assessment of parental report

CONTACTS AND LOCATIONS:
Overall Officials: Kara McNamara, MD, Principal Investigator — ObvioHealth; Vikram Garg, MD, Principal Investigator — Curavit
Locations (1):
- Virtual Site Location - Curavit, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No